CLINICAL TRIAL: NCT07215104
Title: A Prospective Evaluation of Spinal Cord Induced Muscle Stimulation (MuscleSCS) for the Treatment of Chronic Low Back Pain
Acronym: MuscleSCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Francis Hospital (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MuscleSCS Study V2.0
Record Dates: First submitted 2025-10-08; First posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Chronic Low Back Pain (CLBP)

STUDY DESIGN:
Intervention Model Description: The population for this study will include two specific groups of the same pain population. Group one is the Pre-existing SCS Group, these are pain patients with chronic back pain, and who have been implanted with an SCS system with a percutaneous lead or a paddle lead and BurstDRTM IPG for more than 6 month and having success with their BurstSCS stimulation (>50% pain relief).
  Group two is the Trial SCS Group, these are pain patients with chronic back pain, and who have been determined to be candidates for trial and potential permanent SCS with a percutaneous lead or a paddle lead and BurstDRTM IPG.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: MuscleSCS — The population for this study will include two specific groups of the same pain population. Group one is the Pre-existing SCS Group, these are pain patients with chronic back pain, and who have been implanted with an SCS system with a percutaneous lead or a paddle lead and BurstDRTM IPG for more than 6 month and having success with their BurstSCS stimulation (>50% pain relief).
  Group two is the Trial SCS Group, these are pain patients with chronic back pain, and who have been determined to be candidates for trial and potential permanent SCS with a percutaneous lead or a paddle lead and BurstDRTM IPG.

SUMMARY:
This study is a prospective, multi-center study designed to compare the safety and efficacy of spinal cord induced muscle stimulation (MuscleSCS) for the treatment of chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with PSPS type 1 and 2
2. Patients with predominant back pain
3. Patient must be willing and able to provide written informed consent before any clinical investigation-related procedure
4. Age ≥18 y
5. Patients with SCS(BurstDR) stimulation in situ for more than 6 month and >50% pain relief. Patients have to be satisfied with their existing SCS therapy and predominantly use a BurstDR stimulation program.

   (Only responders to that therapy should be included, not patients who have not responded to their therapy so far.) [GROUP 1]
6. Low back pain baseline score of ≥6 on NRS before spinal cord stimulation therapy and a MCID (Minimal clinically important difference) of >50% with SCS(BurstDRTM) trial stimulation. [GROUP 2]
7. Willing and able to comply with the instructions for use, operate the study device, and comply with this clinical investigation plan

Exclusion Criteria:

1. Pathology seen on imaging tests obtained within the past 12 month that is clearly identified and is likely the cause of the CLBP, that can be addressed with surgery
2. Primary symptom of leg pain, or leg pain is greater than back pain
3. Back pain is due to any of the following: vascular causes (eg, aortic aneurysm), spinal infection (eg, osteomyelitis), inflammation or damage to the spinal cord (eg, arachnoiditis or syringomyelia), tumor or spinal metastases
4. Has widespread pain (eg, fibromyalgia) or pain in other area(s), not intended to be treated in this study (eg, neck pain, shoulder pain)
5. Patient has used a morphine equivalent daily dose of >50 MME in the last 30 days
6. Patients with regular intake of systemic steroids (except inhaled steroids used to treat asthma)
7. Imaging (MRI, CT, x-ray) findings within the last 12 mon that contraindicate lead placement
8. Known allergic reaction to implanted materials
9. Severe scoliotic deformity (>11◦ in thoracic or lumbar spine)
10. Patient has a history of or existing intrathecal drug pump
11. Patient with other existing implantable electrical devices, i.e. pacemakers, bladder stimulators, etc.
12. Patient has previous experience with neuromodulation devices, including a failed trial
13. BMI >40
14. Patient is enrolled, or intends to participate, in another clinical drug and/or device study or registry that may interfere with the results of this study.
15. Presence of other anatomic or comorbid conditions, or other medical, social, or psychologic conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements of the clinical investigation results
16. Failed psychologic evaluation
17. Suspicion or evidence of untreated mental illness, substance abuse, or drug-seeking behavior
18. Patient is in current litigation for back pain/injury, or is currently receiving worker's compensation
19. Pregnant or nursing subjects and those who plan pregnancy during the clinical investigation follow-up period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2026-10-07 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
NRS | Enrollment to End of Study (3mo Visit)
  Numerical Rating Scale for Pain
ODI | Enrollment to End of Study (3mo Visit)
  Oswestry Disability Index
EQ5D-5L | Enrollment to End of Study (3mo Visit)
  5 Dimension Health Related Quality of Life Questionnaire
PDI | Enrollment to End of Study (3mo Visit)
  Pain Disability Index
PCS | Enrollment to End of Study (3mo Visit)
  Pain Catastrophizing Scale
PGIC | Enrollment to End of Study (3mo Visit)
  Patient Global Impression of Change

CONTACTS AND LOCATIONS:
Overall Officials: Timothy R Deer, MD, Principal Investigator — WVUM/Thomas Hospitals (Saint Francis Hospital) Spine and Nerve Center
Locations (1):
- WVUM/Thomas Hospitals (Saint Francis Hospital) Spine and Nerve Center, Charleston, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No